CLINICAL TRIAL: NCT02872441
Title: Characterization of Tissular T Follicular Helper Cells in IgG4-RD
Acronym: TIFOLH4
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2016-28; 2016-A00943-48 (Registry Identifier: IDRCB)
Record Dates: First submitted 2016-08-16; First posted 2016-08-19 (Estimated); Last update posted 2023-10-30 (Actual); Status verified 2023-10

CONDITIONS: Disease Immunoglobulin G4
MeSH Terms: interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- diagnosis of disease associated with IgG4 (Experimental): patients suffering from organ initially compatible with a diagnosis of a disease associated with IgG4
  Interventions: Biological: blood sample

INTERVENTIONS:
Biological: blood sample — One blood sample of 50 milliliter 24 hours after the inclusion

SUMMARY:
IgG4-related disease (IgG4-RD) is a recently identified rare disease characterized by inflammatory lesions with polyclonal lymphoplasmocytic infiltrate, with IgG4+ plasma cells predominance, and fibrosis in involved tissues. Despite a preferential involvement of exocrine organs, virtually all tissues can be affected by the disease. Corticosteroids are usually effective in this indication, but with poor tolerance and a high risk of relapse after decrease or withdrawal of this treatment. In this context, identification of new therapeutic targets is a major concern for these patients. Physiopathology of IgG4-RD remains actually unknown. In previous studies, it has been shown that T follicular Helper (Tfh) cells are expanded in the blood of these patients. Tfh cells have an important role in the formation of germinal centers (GCs), and ectopic GCs have been found in tissues of patients with IgG4-RD. Tfh cells have a major role in proliferation and differentiation of B cell compartment. In this context, this population could have an important contribution in the pathophysiology of IgG4-RD and could represent a therapeutic target in this disease.

TIFOLH4 study intend to analyze tissue Tfh cells in patients with IgG4-RD at diagnosis. This study is an exploratory prospective multicentric study. Thirty patients with a suspected diagnosis of IgG4-RD, because of 1 or more suggestive organ involved, will be included in the study. A 50 mL blood sample and a biopsy, obtained in the same time of the diagnostic biopsy sample, will be obtained in this study. The results obtained in patients with a confirmed diagnosis of IgG4-RD (" IgG4-RD group ") will be compared to results of patients with another diagnosis (" control group "). Main objective of the study is to show by confocal microscopy an expansion of the number of Tfh cells (CD3+CD4+PD1+ cells) in tissue of IgG4-RD patients compared to controls. Secondary objectives include : tissue analysis of Tfh subsets (Tfh1, Tfh2 and Tfh17) ; tissue analysis of B regulatory cells, T regulatory cells, and T helper cells (Th1, Th2, Th17); correlation between tissue and circulating biomarkers; tissue proteomic analysis; and functional analysis of circulating Tfh cells after sorting of these cells and co-culture tests with autologous naive B cells. All these results will be compared between the " IgG4-RD group " and the " control group ". This study should clarify the role of these Tfh populations in IgG4-RD, identify diagnostic tissue and blood biomarkers, and identify therapeutic targets in these patients.

ELIGIBILITY:
Inclusion Criteria:

* Patient with a diagnosis of disease associated with IgG4
* Patient signed a consent
* Patient affiliated to the social security scheme

Exclusion Criteria:

* Patients with a corticosteroid therapy current or less than 3 months.
* Patients with an immunosuppressive treatment or being less than 3 months
* Patients with a biotherapy treatment by ongoing or less 6 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2018-02-14 (Actual); Primary Completion 2021-02-08 (Actual); Study Completion 2021-02-08 (Actual)

PRIMARY OUTCOMES:
Location of TFH cells by immunofluorescence technical | 36 months
  Ratio of TFH cell on the number of total T lymphocytes by high power field in confocal microscopy in tissues of patients

CONTACTS AND LOCATIONS:
Locations (1):
- Assistance Publique Hôpitaux de Marseille, Marseille, France

IPD SHARING:
Plan to Share IPD: No